CLINICAL TRIAL: NCT00601809
Title: Gastrografin Use in Small Bowel Obstruction Caused by Adherences
Brief Title: (Gastrografin Use in Small Bowel Obstruction Caused by Adherences)
Acronym: GUSBOCA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Dr. Fausto Catena M.D. PhD, S. Orsola Malpighi University Hospital - University of Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GUSBOCA
Record Dates: First submitted 2008-01-14; First posted 2008-01-28 (Estimated); Last update posted 2008-01-28 (Estimated); Status verified 2008-01

CONDITIONS: Adhesive Small Intestine Obstruction
Keywords: Gastrointestinal; Adhesive Small Intestine Obstruction; Oral water soluble contrast; Non-operative Conservative Management; Operative rate; Hospital stay
MeSH Terms: interventions — Meals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GG (Experimental)
  Interventions: Drug: Gastrografin®: G
- TT (Other)
  Interventions: Other: traditional conservative treatment (TT)

INTERVENTIONS:
Other: traditional conservative treatment (TT) — In the control group (TT: Traditional Treatment), the patients have been treated as in our daily surgical practice of traditional conservative treatment for ASIO, consisting in nil per os diet, nasogastric tube (NGT) decompression and intravenous fluid resuscitation therapy with electrolytes imbalances correction.
  Arms: TT
Drug: Gastrografin®: G — The study group (GG: Gastrografin Group) received, beyond the traditional conservative treatment for ASIO above mentioned, a G meal with a follow-through study immediately.
  Other Names: water-soluble contrast medium (Gastrografin®: G) meal
  Arms: GG

SUMMARY:
Adhesive small intestine obstruction (ASIO) is an important cause of hospital admission and a very common disease. Any improvement in this field will benefit many patients by reducing the operative rate. Patients with this disease are difficult to evaluate and to manage and their treatment is controversial. Emergency surgery is mandatory when strangulation is suspected or in the case of total obstruction. On the other hand, conservative non-operative treatment is indicated in the case of partial obstruction. The role of water-soluble contrast medium (Gastrografin®: GG) in ASIO is still debated with regard to the therapeutic value.

The aim of our study was to determine the therapeutic role of Gastrografin in patients with small intestine obstruction without strangulation caused by adherences (ASIO).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years)
* History of previous abdominal surgical procedures
* Clinical and radiological evidence of adhesive small intestine obstruction without signs of strangulation and peritonism
* ASA I-III patients
* Informed consent

Exclusion Criteria:

* Suspicion of strangulation
* Actual presence or high suspicion of intra-abdominal malignancy
* Suspicion or history of peritoneal carcinomatosis
* active inflammatory bowel disease
* Positive history of radiotherapy on the abdominal region
* Obstructed hernias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2003-09; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
The operative rate in ASIO patients | Within 72 hours and during hospital stay

SECONDARY OUTCOMES:
The incidence of major and minor complications of treatments in the two arm | 1 year
The ASIO recurrences | 1 year
The time to resolution of obstruction | Within hospital stay
The length of hospital stay | Within hospital admission period

CONTACTS AND LOCATIONS:
Overall Officials: Fausto Catena, MD, PhD, Principal Investigator — S.Orsola-Malpighi University Hospital - University of Bologna; Luca Ansaloni, MD, Principal Investigator — S.Orsola-Malpighi University Hospital - University of Bologna; Margherita Gavioli, MD, Principal Investigator — University of Modena and Reggio Emilia; Salomone Di Saverio, M.D., Principal Investigator — S.Orsola-Malpighi University Hospital - University of Bologna
Locations (2):
- Italy (2):
  - S.Orsola-Malpighi University Hospital - University of Bologna, Bologna
  - Emergency Surgery Department - University of Modena, Modena

REFERENCES:
- [Derived] Di Saverio S, Catena F, Ansaloni L, Gavioli M, Valentino M, Pinna AD. Water-soluble contrast medium (gastrografin) value in adhesive small intestine obstruction (ASIO): a prospective, randomized, controlled, clinical trial. World J Surg. 2008 Oct;32(10):2293-304. doi: 10.1007/s00268-008-9694-6. PMID 18688562